CLINICAL TRIAL: NCT05137431
Title: Comparison of High-flow Nasal Oxygenation and Non-invasive Ventilation Strategies for the Treatment of Covid-19 Pneumonia in the Intensive Care Unit: a Prospective Trial.
Brief Title: High-flow Nasal Oxygenation and Non-invasive Ventilation Strategies for the Treatment of Covid-19 Pneumonia
Status: Completed | Type: Observational
Sponsor: Medipol University (Other)
Responsible Party: Principal Investigator, Bahadir Ciftci, Primary researcher, Medipol University
Other Study IDs: Medipol Hospital 22
Record Dates: First submitted 2021-11-26; First posted 2021-11-30 (Actual); Last update posted 2022-08-11 (Actual); Status verified 2022-08

CONDITIONS: COVID-19 Pneumonia; COVID-19 Acute Respiratory Distress Syndrome
MeSH Terms: interventions — Noninvasive Ventilation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- High Flow Nasal Oxygenation-HFNO: The current will be adjusted from 50-70 liters. The patient's SpO2 value will be maintained at at least 92%. Arterial blood gas will be checked at the 1st hour
  Interventions: Other: HFNO and NIV
- Non-Invasive Ventilation-NIV: Tidal volume will be adjusted to be 6-8 ml/kg. The respiratory rate will be <30. The patient's SpO2 value will be maintained at at least 92%. The PEEP value will be 5 cmH2O. At the 1st hour, arterial blood gas will be checked.
  Interventions: Other: HFNO and NIV

INTERVENTIONS:
Other: HFNO and NIV — Patients meeting the inclusion criteria will be treated alternately with 2 hours of HFNO and 1 hour of NIV (HFNO-NIV for the same patient in turn). In 24 hours, there will be 16 hours of HFNO, 8 hours of NIV.
  Parameters to record
  * Respiratory parameters (respiratory rate)
  * SpO2
  * Ventilator settings
  * Patient's tolerance (VAS; between 0-100)
  * Arterial blood gas (HFNO and NIV at 1 hour)
  * Clinical parameters (D dimer, CRP, ROX index)
  Intubation criteria
  * Loss of consciousness
  * Agitation
  * Persistent hypotension
  * Need for fluid resuscitation
  * Need for vasopressor
  * Respiration rate ≥40/min
  * SpO2 <92
  * pH<7.30

SUMMARY:
HFNO and NIV strategies are the most commonly used strategies for the treatment of hypoxia in patients with a diagnosis of COVID-19 who are still followed in the intensive care unit, but there is no study comparing the two yet. In our prospective study, we aimed to compare these two treatment modalities. The primary goal is that the treatment is successful (weaned off HFNO/weaned off NIV: No need for HFNO or NIV and the patient recovers without the need for intubation). Failure will be evaluated as the need for intubation during treatment or the patient's death. Secondary aim is failure of treatment and discharge of patients from intensive care to service or home.

DETAILED DESCRIPTION:
Coronavirus 2019 disease (COVID-19) is a deadly infection that causes a new type of severe acute respiratory syndrome. It has been reported that the mortality rate in critically ill patients with a diagnosis of COVID-19 reached 61%. The primary pathology in these patients is progressive hypoxia due to lung injury and associated multi-organ damage. It has been reported that aggressive treatments such as tracheal intubation and classical mechanical ventilation to treat lung injury are not helpful or even harmful. The highest mortality rate was reported as 86% in these patients on mechanical ventilation. Acute respiratory distress syndrome (ARDS) developing in COVID-19 infection is not typical and is estimated to have a different mechanism, therefore it is emphasized that different strategies should be used for the treatment of ARDS in these patients. Two of the most important strategies used in these patients followed in the intensive care unit are high flow nasal oxygenation (High Flow Nasal Oxygenation-HFNO) and non-invasive ventilation (Non-Invasive Ventilation-NIV). HFNO is a method frequently used before intubation in adult patients with acute respiratory failure. It is based on the principle of giving warm and humidified oxygen to the patient through a nasal cannula in the range of 1-70 L/min. Due to the low number of mechanical ventilators in many intensive care units at the beginning of the pandemic, it was used in many COVID-19 patients and was found to be effective in later retrospective analyzes. It has been reported in many studies that HFNO therapy is more effective than conventional mask oxygen therapy. There are publications stating that it is more advantageous compared to NIV as it is easier to apply and more comfortable for the patient. Conventional NIV is called continuous positive airway pressure (CPAP) or Bi-level positive airway pressure (BiPAP) ventilation. It is used as oxygen/ventilation therapy in SARS and H1N1 patients. Studies have reported that it is used in 70% of patients before tracheal intubation in COVID-19 patients. However, mortality was high in these patients.

HFNO and NIV strategies are the most commonly used strategies for the treatment of hypoxia in patients with a diagnosis of COVID-19 who are still followed in the intensive care unit, but there is no study comparing the two yet. In our prospective study, we aimed to compare these two treatment modalities. The primary goal is that the treatment is successful (weaned off HFNO/weaned off NIV: No need for HFNO or NIV and the patient recovers without the need for intubation). Failure will be evaluated as the need for intubation during treatment or the patient's death. Secondary aim is failure of treatment and discharge of patients from intensive care to service or home.

ELIGIBILITY:
Inclusion Criteria:

* PCR (+)
* P/F ≤300 mmHg (despite standard mask oxygen support from 15 L/min for 15 minutes)
* Respiratory rate ≥24/min or signs of respiratory failure (intercostal retraction, nasal wing breathing)

Exclusion Criteria:

* Chronic respiratory failure
* Cardiogenic pulmonary edema
* Aplasia
* GCS ≤12
* Hemodynamic instability (use of vasopressors)
* Emergency intubation requirement

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: This prospective, single-center study will be conducted in the Intensive Care Unit of Medipol Mega Hospital, an academic university hospital. It is planned to include patients over the age of 18 with a diagnosis of COVID 19 (severe respiratory failure and positive PCR test).
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2021-12-08 (Actual); Primary Completion 2022-04-30 (Actual); Study Completion 2022-04-30 (Actual)

PRIMARY OUTCOMES:
Success of the treatment | Through study completion, an average of 2 months
  The primary goal is that the treatment is successful (weaned off HFNO/weaned off NIV: No need for HFNO or NIV and the patient recovers without the need for intubation).

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul Medipol University Hospital, Istanbul, Bagcilar, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
We will not plan to share IPD

REFERENCES:
- [Background] Calligaro GL, Lalla U, Audley G, Gina P, Miller MG, Mendelson M, Dlamini S, Wasserman S, Meintjes G, Peter J, Levin D, Dave JA, Ntusi N, Meier S, Little F, Moodley DL, Louw EH, Nortje A, Parker A, Taljaard JJ, Allwood BW, Dheda K, Koegelenberg CFN. The utility of high-flow nasal oxygen for severe COVID-19 pneumonia in a resource-constrained setting: A multi-centre prospective observational study. EClinicalMedicine. 2020 Nov;28:100570. doi: 10.1016/j.eclinm.2020.100570. Epub 2020 Oct 6. PMID 33043285
- [Background] Frat JP, Brugiere B, Ragot S, Chatellier D, Veinstein A, Goudet V, Coudroy R, Petitpas F, Robert R, Thille AW, Girault C. Sequential application of oxygen therapy via high-flow nasal cannula and noninvasive ventilation in acute respiratory failure: an observational pilot study. Respir Care. 2015 Feb;60(2):170-8. doi: 10.4187/respcare.03075. Epub 2014 Oct 7. PMID 25294935